CLINICAL TRIAL: NCT04471610
Title: Point Of Care With Serial NT-proBNP Measurement in Patients With Acute Decompensation of Heart Failure as a Therapy-monitoring During Hospitalization: A Prospective, Unblinded, Randomized, Controlled Pilot Trial - The POC-HF Trial
Brief Title: Point Of Care With Serial NT-proBNP Measurement in Patients With Acute Decompensation of Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Professor of Internal Medicine, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-01030
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Potassium; Sodium

STUDY DESIGN:
Intervention Model Description: In the intervention arm serial measurement of NT-proBNP will be made available to the treating physician. A control group continuing to undergo care according to the 2016 ESC Guidelines will serve as comparator. Changes in NT-proBNP levels, safety laboratory parameters such as sodium, potassium, creatinine, HF medication, vital signs, body weight and BMI, QoL, length of hospital stay, NYHA functional class, adverse events, transfer to the Intensive Care Unit and mortality will be recorded in patients with ADHF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group A: Patients allocated to the control group will undergo the measurements at inclusion and discharge visit. The control group conduces to compare the NT-proBNP and HF medication changes under therapy monitoring with serial NT-proBNP measurements to the NT-proBNP and HF medication changes with sign and symptom guided HF therapy. The diagnostic and therapeutic decisions in the control Group and in the Intervention group will be based on the current 2016 ESC guidelines on the diagnosis and therapy of HF as established at the KSBL Liestal. At discharge, the same measurements as at the inclusion visit will be repeated in all patients to monitor the effects associated with the participation in this trial.
- POC-available group (Experimental): Group B:Patients allocated to the intervention group (POC-available group) will undergo serial measurements of NT-pro BNP, potassium, sodium, and creatinine every second business day. The blood collection (10 ml of Lithium Heparin blood) for these tests will be done in the morning together with the regularly blood collection. The study team does the the analysis on the study devices. The result of the test will be provided directly to the responsible physician. Treatment changes are at the discretion of the responsible physician. The physician will be alerted by a phone call of a study member if the NT-proBNP hasn't decreased by 10% or more between two measurements. But no specific recommendations with regards to therapy will be provided by the investigator or his team. However, diagnostic and therapeutic decisions will be based on the current 2016 ESC guidelines on the diagnosis and therapy of HF as established at the KSBL Liestal.
  Interventions: Other: Serial measurements of NT-pro BNP, potassium, sodium, and creatinine every second business day

INTERVENTIONS:
Other: Serial measurements of NT-pro BNP, potassium, sodium, and creatinine every second business day — Serial measurements of NT-proBNP, sodium, potassium, and creatinine in the NT-proBNP-group vs. no serial measurements in control group. In the intervention group the body weight, vital parameters, therapy changes and adverse events are documented the above mention serial measurement every second business day.
  Arms: POC-available group

SUMMARY:
The goal of this study is to explore whether the availability of serial NT-proBNP measurements together with safety parameters such as electrolytes and creatinine may influence treatment decision in patients with acute decompensated heart failure (ADHF) leading to more rapid and faster dose increase of prognostic therapies and earlier hospital discharge.

DETAILED DESCRIPTION:
The proposed study is a prospective, unblinded, single center, 2-arm randomized controlled pilot trial. In the intervention arm serial measurement of NT-proBNP will be made available to the treating physician. A control group continuing to undergo care according to the 2016 ESC Guidelines will serve as comparator. Changes in NT-proBNP levels, safety laboratory parameters such as sodium, potassium, creatinine, Heart failure (HF) medication, vital signs, body weight and BMI, Quality of Life (QoL), length of hospital stay, New York Heart Association (NYHA) functional class, adverse events, transfer to the Intensive Care Unit and mortality will be recorded in patients with ADHF.

The Kantonsspital Baselland (KSBL) Liestal will be the only study center. All members of the study group will the thoroughly instructed regarding study procedures. Inclusion visits will be conducted only by a member of the study group. All Patients with ADHF on the medical ward of the KSBL Liestal will be provided an information sheet regarding goals and procedures of the study and the informed consent. Inclusion criteria will be checked after admission. Patients not matching the inclusion criteria at the screening visit cannot participate in this study. Patients will be provided sufficient time for their decision. The investigators communicate clearly that participation in the study is absolutely voluntary and refusal of participation has no influence on treatment during hospitalization.

In order to minimize bias that may be introduced by even minor differences in executing and interpreting technical exams, all study related measurements and procedures will be performed in a centralized manner at the KSBL Liestal.

Patients will be included only after approval of informed consent. Randomization is performed using 50 closed envelopes containing a paper shit with either the letter A or B. In total there are 25 A's and 25 B's. The letter A stands for the control group and the letter B for the intervention group. These envelopes are mixed initially, numbered for order purposes and the order maintained throughout the study. The name of the patient will be written down on the envelope. Then it will be open and the patient will be allocated to the study group depending on the letter in the envelope. All patients will undergo an inclusion and discharge visit. General demographic data, including age, gender, nationality, smoking status, alcohol consumption, current profession, exercise behavior, allergies, medication, HF history and comorbidities will be recorded. Assessment of vital signs and body weight will be performed together with an electrocardiogram, several laboratory tests (NT-proBNP, potassium, sodium and creatinine). In addition, questionnaires concerning QoL (SF-12, KCCQ, MLWHFQ) will be filled in by the participants. Women who can get pregnant (not yet in menopause and last menstrual period less than 12 months, not surgically sterilized, ovaries and/or uterus not removed) will have to undergo a pregnancy test prior to inclusion into the study.

Patients allocated to the intervention group (POC-available group) will undergo serial measurements of NT-pro BNP, potassium, sodium, and creatinine every second business day. The investigators have chosen this time-lag because an earlier time point would not show the change of the security parameter creatinine due to longer half-life-time. For this test, blood is collected from the patients. These samplings will be done in the morning together with the regularly blood collection through the attending nurse according to the established procedure of the KSBL Liestal in the morning. 10ml blood will be collected for this study during each blood sample with a standard Lithium-blood-collection tube. Members of the study team will collect the blood samples and analyses them on the study devices. The result of the test will be provided directly to the responsible physician of the medical department at the KSBL Liestal. Treatment changes are at the discretion of the responsible physician. The physician will be alerted by a phone call of a study member if the NT-proBNP hasn't decreased by 10% or more between two measurements. But no specific recommendations with regards to therapy will be provided by the investigator or his team. However, diagnostic and therapeutic decisions will be based on the current 2016 ESC guidelines on the diagnosis and therapy of HF as established at the KSBL Liestal.

Patients allocated to the control group will undergo the measurements at inclusion and discharge visit. The control group conduces to compare the NT-proBNP and HF medication changes under therapy monitoring with serial NT-proBNP measurements to the NT-proBNP and HF medication changes with sign and symptom guided HF therapy. As in the intervention group, diagnostic and therapeutic decisions in the control group will be based on the current 2016 ESC guidelines on the diagnosis and therapy of HF as established at the KSBL Liestal. At discharge, the same measurements as at the inclusion visit will be repeated in all patients to monitor the effects associated with the participation in this trial.

Total study duration will cover a period of approximately 3 years. Patients will be screened until a total of 25 patients are included per study group.

Overall, 50 patients are planned to be recruited. Recruitment is estimated to start in September 2017 and end at the latest in March 2020 after discharge of the last hospitalized patient included in the study. Data collection of the study is expected to be completed by May 2020 and data analysis by December 2020.

The expected duration of the study for each patient will be defined by the time period from inclusion to discharge and is expected to be in the range of 8-12 days (=average time for HF hospitalization of our institution).

As an university institution, the KSBL Liestal mandates its physician and nursing staff to provide evidence-based medical care and to follow recognized and established national and/or international guidelines whenever possible. Nevertheless, deviation from guidelines may be necessary in specific cases. The decision whether and when to deviate from guidelines is at the discretion of the responsible physician and nursing staff and is taken to the best individual knowledge. Patients with ADHF admitted to the Intensive Care Unit are not included in this study. Patients not requiring intensive care treatment will be hospitalized on a regular medical ward and treated with diuretics to improve symptoms of congestion. In case a patient is transferred to the Intensive Care Unit after study inclusion, further data from date of transfer onwards will not be collected, to avoid discomfort to patients and medical personal while the patient is in a critical situation. The study itself is also composed for treatments on a regular medical ward. The transfer to the Intensive Care Unit will serve as the endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* NYHA functional class II or III
* Symptoms of heart failure:

E.g.: Dyspnea Paroxysmal nocturnal dyspnea Reduced exercise capacity Fatigue Extended recovery after exercising Peripheral edema (lower leg, ankle) NT-proBNP >300 (pg/ml)

* Age > 18 Years

Exclusion Criteria:

* NYHA functional class I or IV
* NT-proBNP < 1200 pg/ml and creatinine clearance < 60 ml/min (Clearance (ml/min) = 1.23(women 1.03) x body weight (Kg) x (140-Age)/ creatinine (umol/L)) Creatinine clearence: ___________ <60ml/min
* Heart failure due to chemotherapeutic drugs
* Uncontrolled brady- or tachyarrythmia
* Unstable angina pectoris
* Severe uncorrected valvular disease
* Planned cardiac intervention in the next 6 months
* Clinically significant concomitant disease states:

On-going cancer treatment

* Active infection
* Immunosuppressive medical therapy
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the study procedures (Due to language problems, psychological disorders, dementia, etc.)
* Participation in another intervention study
* Enrolment of investigators or their family members
* Pregnancy, lactation, breast feeding
* Positive pregnancy test for females in childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Changes in NT-proBNP | Up to 4 weeks, on average 10 days
  Meassurement of NT-proBNP
Dosage and variations in medication to treat heart failure | Up to 4 weeks, on average 10 days
  Changes in medical heart failure therapies such as Diuretics, Nitrates, Angiotensin-converting-enzyme (ACE) Inhibitors or angiotensin-receptor blockers (ARBs), Beta blocker

SECONDARY OUTCOMES:
HR (in beats/min) | Up to 4 weeks, on average 10 days
  Vital signs
BP (in mmHg) | Through study completion, on average 10 days
  Vital sign
BMI and Body weight | Up to 4 weeks, on average 10 days
  Body mass index and weight in kg
KCCQ (Kansas City Cardiomyopathy ) Questionnaire | Up to 4 weeks, on average 10 days
  The KCCQ is a self-administered, 23-item questionnaire measuring HRQoL in patients with CHF regardless of its origin. Each item has a 5-, 6-, or 7-point Likert scale. The questionnaire assesses six domains of HRQoL: Physical Limitation, Symptoms, Symptom Stability, Social Limitation, Self-Efficacy, and Quality of Life. Domain scores were transformed to 0-100 (highest level of functioning) scales.
SF12 (Short Form 12 Health Survey ) Questionnaire | Up to 4 weeks, on average 10 days
  A mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Minnesota LIVING WITH HEART FAILURE® Questionnaire | Up to 4 weeks, on average 10 days
  The questionnaire is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses.
  The instrument can be used as a key outcome measure in studies and evaluations of outpatients with symptomatic (NYHA class II to IV) heart failure with a reduced or preserved ejection fraction. This patient-reported outcome can be used to determine whether a treatment for heart failure is effective for improving patients' quality of life by reducing the adverse impact of heart failure.
Potassium | Up to 4 weeks, on average 10 days
  Meassurement of potassium as safety parameter
Sodium | Up to 4 weeks, on average 10 days
  Meassurement of sodium as safety parameter
Creatinine | Up to 4 weeks, on average 10 days
  Meassurement of creatinine as safety parameter
Length of hospital stay | Up to 4 weeks, on average 10 days
  Days spent in the hospital
NYHA functional class | Up to 4 weeks, on average 10 days
  NYHA class I-IV
Transfer to the Intensive Care Unit (ICU) | Number pf patients
  Stay at ICU

CONTACTS AND LOCATIONS:
Overall Officials: Jörg D. Leuppi, Prof., Principal Investigator — Head of Medical University Clinic, Cantonal hospital Baselland
Locations (1):
- Cantonal Hospital Baselland Liestal, Liestal, Basel-Landschaft, Switzerland